CLINICAL TRIAL: NCT05691556
Title: Study of the Sensitivity to Change of a Bimanual 3D Analysis Protocol for the Assessment of Upper Limb Movement in Children With Cerebral Palsy Before and After Therapies
Acronym: BE API CHANGE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC21.0299 - BE API CHANGE
Record Dates: First submitted 2023-01-02; First posted 2023-01-20 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Cerebral Palsy Infantile
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Children CP: Children with cerebral palsy with motor impairment of the upper limb(s), seen in consultation and included in a HABIT-ILE therapeutic program and/or botulinum toxin injections
  Interventions: Procedure: HABIT ILE rehabilitation course; Procedure: botulinum toxin injections

INTERVENTIONS:
Procedure: HABIT ILE rehabilitation course — The HABIT-ILE course, created by the Belgian team of Prof. Yannick Bleyenheuft, is a rehabilitation of the upper and lower limbs, following the concepts of structured motor learning and intensive therapy. The internships last 2 weeks and are performed on a multi-year basis since 2018 at the SSR pediatric, Fondation Ildys, Site de Ty Yann in Brest.
  In this group, upper limb assessments are performed the week before and the week after the HABIT ILE training course
Procedure: botulinum toxin injections — Toxin injections are used for their effect on the local reduction of spasticity after intramuscular injection. This treatment is usually offered to these children every 6 months or so for functional improvement.
  These botulinum toxin injections are organized on a weekly basis in a pediatric day hospital (CHU Morvan in Brest).
  In this group, upper limb assessments were performed 0-2 weeks before and then 4 to 6 weeks after the botulinum toxin injections (see table below), at the peak of the toxin's efficacy.

SUMMARY:
Cerebral Palsy is the most common cause of motor disability in children. It can lead to a deficit of the upper limb which alters the realization of daily activities, in particular in bimanual situations, and eventually leads to a decrease in their participation.

Three-dimensional (3D) movement analysis is a tool that provides an accurate and objective measurement of movement. This technology allows us to understand and characterize movement anomalies in order to guide and adapt therapies to the upper limb. The majority of 3D upper limb analysis protocols used to measure the effect of interventions, such as botulinum toxin injections indicated for the treatment of spasticity or other innovative rehabilitative therapies, are unimanual and do not study bimanual function, which is more representative of the actual use of the upper limbs in daily life.

Recently, a 3D bimanual analysis protocol called "Be An Airplane Pilot" (BE-API), taking place in an innovative play context, has been developed and validated in PC children. The 2nd version of the protocol (BE API 2.0) also allowed the exploration of new parameters in a bimanual situation such as the fluidity and the trajectory of the movement. In order to determine the interest of the BE API 2.0 protocol in routine clinical evaluation of the upper limbs, its sensitivity to change, i.e. its capacity to detect modifications caused by a therapy on the movements of the upper limbs is necessary (e.g.: Hand and Arm Bimanual Intensive Therapy Including Lower Extremity (HABIT ILE), botulinum toxin injections).

ELIGIBILITY:
Inclusion Criteria:

* Child between the ages of 5 and 18,
* Child with cerebral palsy as defined by the CSEP
* Level of manipulation sufficient to perform the tasks of the 3D protocol (MACS score I to III included),
* For whom the HABIT-ILE therapeutic program and/or botulinum toxin injection is prescribed
* Affiliated via his/her parents to a social security plan,
* No opposition formulated by the holders of parental authority and the child

Exclusion Criteria:

* Child with unilateral or bilateral spastic cerebral palsy
* Cognitive deficits hindering the comprehension of instructions or visual disorders not allowing the visualization of the game board,
* Pain in the upper limb (VAS score>3),
* Contraindications to the use of botulinum toxins and absence of indications as mentioned in the HAS 2010 recommendations
* Patients under legal protection (guardianship, curatorship, ...)
* Refusal to participate

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children with cerebral palsy with motor impairment of the upper limb(s), seen in consultation and included in a HABIT-ILE therapeutic program and/or botulinum toxin injections.
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2020-07-16 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
To study the sensitivity to change of the BE API 2.0 bimanual 3D analysis protocol by measuring the change in the severity of movement deviation in the upper limb before and after therapy | 2 months
  The Arm Profile score is a kinematic index that reflects the severity of the subject's movement deviation compared to the "normal" deviation of healthy children.

SECONDARY OUTCOMES:
To measure the change induced by the therapy on the parameters measured in movement analysis (kinematic), clinical and functional measures at the deficient MS (comparison before and after therapy). | 2 months
  kinematic parameters measured in motion analysis with the BE API 2.0 protocol
To measure the change induced by the therapy on the parameters measured in movement analysis (spatio-temporal), clinical and functional measures at the deficient MS (comparison before and after therapy). | 2 months
  Spatio-temporal parameters measured in motion analysis with the BE API 2.0 protocol
To study the association between the parameters measured in motion analysis clinical/functional measurements (kinematics and spatio-temporal parameters) before and after therapy. | 2 months
  Correlation of motion analysis measurements (kinematics and spatio-temporal parameters) measured with the BE API 2.0 protocol before and after therapy to clinical.
To study the association between the parameters measured in motion analysis with the BE API 2.0 protocol (kinematics and spatio-temporal parameters) before and after therapy. | 2 months
  Correlation of motion analysis measurements (kinematics and spatio-temporal parameters) measured with the BE API 2.0 protocol before and after functional measurements
Compare the dominant and non-dominant upper limb of PC children on parameters measured in motion analysis with the BE API 2.0 protocol (kinematic and spatio-temporal), before and after therapy. | 2 months
  Compare motion analysis measurements (kinematics and spatiotemporal parameters) of dominant and non-dominant MS measured with the BE API 2.0 protocol before and after therapy

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement.